CLINICAL TRIAL: NCT03674593
Title: Clinical and Fundamental Aspects of Prosthetics and Translocation of Mitral Valve Chordae
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Tomsk National Research Medical Center of the Russian Academy of Sciences (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Mitral Valve Chordae
Record Dates: First submitted 2018-07-09; First posted 2018-09-17 (Actual); Last update posted 2025-04-09 (Actual); Status verified 2025-04

CONDITIONS: Degenerative Mitral Valve Disease
Keywords: Mitral Valve Chordae; Degenerative Mitral Valve Disease; Mitral Valve Chordae Replacement; Mitral Valve Chordae Translocation; Mitral Valve Chordae Prosthetics

STUDY DESIGN:
Intervention Model Description: Single-center, prospective, semi-open, randomized study
Who Masked: Participant
Masking Description: Single blind masking (Participant)
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Mitral valve chordae prosthesis (Experimental): Patients of this group receive mitral valve chordae replacement performed in five stages:
  1. Measure the required length of the chordae.
  2. Forming loops.
  3. Fixation of the loop group to the papillary muscles.
  4. Fixation of chordal loops to the free edge of the valve.
  5. Annuloplasty with a support ring and a hydraulic test to confirm the absence of prolapse.
  Interventions: Procedure: Mitral valve chordae prosthesis
- Mitral valve chordae translocation (Active Comparator): The technique of translocation of secondary chordae:
  The method consists essentially of three stages:
  1. Selection of the secondary chordae.
  2. Fixation of secondary chordae to the free edge of the valve.
  3. Annuloplasty support ring and hydraulic test to confirm the absence of prolapse.
  Interventions: Procedure: Mitral valve chordae translocation

INTERVENTIONS:
Procedure: Mitral valve chordae prosthesis — The method consists of five stages:
  1. Measure the required length of the chords
  2. Forming loops
  3. Fixation of the loop group to the papillary muscles
  4. Fixation of chordal loops to the free edge of the valve
  5. Annuloplasty with a support ring and a hydraulic test to confirm the absence of prolapse
  Other Names: Chordae prosthesis
  Arms: Mitral valve chordae prosthesis
Procedure: Mitral valve chordae translocation — The method consists essentially of three stages:
  1. Selection of the secondary chord.
  2. Fixation of secondary chords to the free edge of the valve.
  3. Annuloplasty support ring and hydraulic test to confirm the absence of prolapse.
  Other Names: Chordae translocation
  Arms: Mitral valve chordae translocation

SUMMARY:
The study compares the efficacies of two surgical procedures for the treatment of mitral valve prolapse due to myxomatous degeneration of the mitral valve: the chordae replacement and the translocation of secondary mitral valve chordae.

DETAILED DESCRIPTION:
Summary: This study compares the efficacy and the safety of two surgical procedures for the treatment of mitral valve prolapse due to degeneration of the mitral valve: chordae replacement and the translocation of secondary mitral valve chordae.

In our study, researchers used the loop method proposed by von Oppel and Mohr in 2000. The main principle of the method of prosthetic chordae is the preservation of the native anatomy of the mitral valve. This principle is achieved by the implantation of artificial chordae made of ePTFE Gore-Tex threads.

The chordae replacement method essentially involves five stages:

1. Measuring the required length of the chordae.
2. Forming the loops.
3. Fixation of the group of loops to the papillary muscles.
4. Fixation of the chordal loops to the free edge of the valve.
5. Annuloplasty with a support ring and a hydraulic test to confirm the absence of prolapse.

Chordae translocation is the alternative method, which does not require measurement and selection of chordae lengths. Chordae replacement is technically easier (less aortic clamping time) with comparable results.

The technique of translocation of secondary chordae essentially consists of three stages:

1. Selection of the secondary chordae.
2. Fixation of secondary chordae to the free edge of the valve.
3. Annuloplasty support ring and hydraulic test to confirm the absence of prolapse.

ELIGIBILITY:
Inclusion Criteria:

1. Isolated type II mitral valve insufficiency by A. Carpentier
2. Mitral regurgitation degree >2
3. Age >18 years
4. Signed informed consent to participate in the study

Exclusion Criteria:

1. Any other cardiac surgeries
2. Age <18 years
3. Multiple organ failure
4. ReDo procedure
5. Persistent atrial fibrillation
6. Acute infective endocarditis
7. Refusal to sign informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 64 (Actual)
Dates: Start 2018-07-09 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Mitral regurgitation degree measure | Two weeks
  Mitral regurgitation degree (from 1 to 4) assessed by echocardiography two weeks after surgery

SECONDARY OUTCOMES:
Surgical efficacy measure | One year
  Mitral regurgitation degree (from 1 to 4) assessed by echocardiography one year after surgery
ERO measure | Two weeks
  Effective regurgitant orifice (ERO) (in square millimeters) assessed by echocardiography two weeks after surgery

CONTACTS AND LOCATIONS:
Overall Officials: Elena N. Pavlyukova, MD, PhD, Principal Investigator — Tomsk NRMC
Locations (1):
- Cardiology Research Institute, Tomsk NRMC, Tomsk, Russia

IPD SHARING:
Plan to Share IPD: No